CLINICAL TRIAL: NCT07210879
Title: Early Predictors for Neurological Outcome After Traumatic Spinal Cord Injury
Acronym: MurnauMAP
Status: Active, not recruiting | Type: Observational
Sponsor: BG Unfallklinik Murnau (Other)
Collaborators: Foundation Wings For Life (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Iris Leister, Head of Research SCI, BG Unfallklinik Murnau
Other Study IDs: 22057
Record Dates: First submitted 2025-09-30; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Acute Traumatic Spinal Cord Injury
Keywords: Spinal cord injuries; Blood pressure; Hemodynamics; Critical care; Biomarkers; Neurological recovery
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- MAP cohort: AIM 1 is to investigate if continuous monitoring of arterial pressure and augmentation via administration of vasopressors during the ICU stay affect the neurological outcome after traumatic SCI.
  For this, data of 161 patients who underwent hemodynamic monitoring in the acute stage after traumatic SCI have been included in the analysis.
- Biomarker Cohort: AIM 3 is to evaluate if diagnostic and/or prognostic biomarkers can be derived from measurements in clinical routine.
  For this analysis, we will include data from 747 patients who had at least five blood samples collected within the first year after injury, with the first sample obtained within two weeks post-injury, and who completed both acute and chronic neurological assessments.
- Opioid Cohort: AIM 2 is to evaluate if other pharmacological interventions - specifically opioids - during the ICU stay are related to neurological recovery after SCI.
  For this, we will analyze data from approximately 240 individuals treated in our ICU who received opioid therapy, including detailed information on timing, dosage, and duration of administration, in relation to their acute and long-term neurological outcomes.

SUMMARY:
This project investigates early predictors of neurological recovery after traumatic spinal cord injury through three main aims:

1. MAP and vasopressors - determine whether continuous monitoring of mean arterial pressure (MAP) and the use of vasopressors in the ICU influence neurological outcome.
2. Pharmacological interventions - evaluate the impact of other medications, particularly opioids in the acute stage, on recovery.
3. Biomarkers - identify diagnostic and prognostic biomarkers (blood-borne or digital) from routine clinical measurements within the first year after injury.

Using high-frequency ICU data and advanced data science methods, the study seeks to provide insights that support individualized treatment strategies and improve outcomes after SCI.

DETAILED DESCRIPTION:
Study rationale In order to address the question whether MAP targets and pharmacological interventions affect the neurological outcome after traumatic SCI, a large sample size of longitudinal data is required. The BG Trauma Center Murnau is a level Ia trauma center in Bavaria (Germany) and approximately 120 patients are treated with acute traumatic SCI every year. Therefore the spinal cord injury center at the Trauma Center Murnau represents one of the largest centers in Europe specializing in the treatment of SCI.

A retrospective analysis of routinely collected data during the ICU stay would create an opportunity to investigate the relation of hemodynamic parameters, pharmacological interventions, and neurological recovery in a large cohort of individuals who sustained acute traumatic SCI.

A better understanding of the effect of interventions in the very acute stages of SCI on neurological recovery, as well as the identification of new biomarkers would be of utmost interest for physicians. The knowledge gain from this study could inform clinical decision-making in the future and would therefore ultimately improve the treatment of acute SCI.

Specific aims and hypothesis of the project:

AIM 1 Investigate if continuous monitoring of arterial pressure and augmentation via administration of vasopressors during the ICU stay affect the neurological outcome in individuals who sustained traumatic SCI.

Hypothesis 1.1 The administration of high doses of vasopressor medication within the acute stage of SCI negatively affects long-term neurological outcome.

Hypothesis 1.2 MAP goals need to be defined depending on several contributing factors, such as the patient's age, the presence of co-morbidities, and medication intake prior to the SCI instead of universal MAP targets for the whole SCI population.

AIM 2 Evaluate if other pharmacological interventions (opioids, sedatives, neuroleptics, pain medication especially neuropathic pain medication) during ICU stay are related to neurological recovery and adverse events after SCI.

Hypothesis Administration of high doses of opioids and sedatives negatively affect the neurological outcome after SCI.

AIM 3 Evaluate if diagnostic (for the presence and severity of SCI), and/or prognostic (for neurological recovery and disease progression) biomarkers (blood-borne, or digital) can be identified derived from routine clinical measurements during the first year after injury in clinical routine in the very acute post-injury phase.

Hypothesis 3 Biomarkers with either a diagnostic value (for injury severity) as well as prognostic markers (for neurological recovery and disease progression) could assist clinical decision-making and would therefore be of utmost interest for treating physicians, and for clinical research.

Detailed research plan:

We will retrospectively analyze routinely collected data from patients who sustained traumatic SCI, and were treated in the ICU at the Trauma Center Murnau (Germany). Data to be extracted from the patient data management system include medication (timing, dosage and cumulative dose), routine blood chemistry data, high frequency hemodynamic parameters, ventilation (duration and technique), and complications (infections, etc.) during the ICU stay. In the first step, we aim to investigate the effect of MAP monitoring, vasopressor administration, and other pharmacological interventions on neurological recovery. In a second step of analysis, we will evaluate if new biomarkers can be derived from routinely collected data. We anticipate that a better understanding of the relation between early interventions during intensive care and neurological recovery, as well as the identification of new biomarkers will inform clinical decision-making in the future and would therefore ultimately improve the treatment of acute SCI.

ELIGIBILITY:
General Inclusion Criteria:

Data from patients who sustained traumatic SCI, and who

* completed at least one neurological examination in the acute / sub-acute stage of injury (between the day of injury and 40 days post-SCI) and in the chronic stage of injury (the latest neurological assessment between day 70 and day 546 after SCI)
* agreed to provide their medical data for research purposes in the European Multicenter Study about Spinal Cord Injury (EMSCI) database

specific for Cohort 1: MAP Cohort patients who

* were initially admitted to the BG Trauma Center Murnau, or transferred for acute SCI care within two days after trauma
* were treated in the intensive care unit (ICU) and underwent hemodynamic monitoring for at least 24 hours

specific for Cohort 2: Biomarker Cohort - patients who had at least five blood samples collected within the first year after injury, with the first sample obtained within two weeks post-injury

specific for Cohort 3: Opioid Cohort

- patients who were treated in the ICU and received opioid therapy, including detailed information on timing, dosage, and duration of administration

Exclusion Criteria:

* Patients with non-traumatic spinal cord injury or non-spinal cord injury
* Patients who were initially admitted and/or surgically treated in another hospital and transferred to the BG Trauma Center Murnau later than two days post-SCI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with traumatic spinal cord injury
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
ISNCSCI | Days after Injury (DAI) 1-546
  International Standards for Neurological Classification about Spinal Cord Injury

CONTACTS AND LOCATIONS:
Locations (1):
- BG Trauma Center Murnau, Murnau am Staffelsee, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.wingsforlife.com/de/forschung/fruehzeitige-vorhersageparameter-neurologischer-erholung-5326